CLINICAL TRIAL: NCT00129454
Title: Telemedicine Treatment for Veterans With Gulf War Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Purpose: Other
Other Study IDs: GWI 04-355
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Gulf War Syndrome
Keywords: Telemedicine; Cognitive Behavior Therapy; Utilization; Randomized Control Trial; Gulf War Illness; Symptom-Based Illness; Multisymptom Illness; High utilization
MeSH Terms: conditions — Persian Gulf Syndrome; Patient Acceptance of Health Care | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telemedicine treatment (Experimental): Psychotherapy delivered by telephone
  Interventions: Behavioral: Cognitive Behavioral Therapy
- In-Person treatment (Active Comparator): Psychotherapy delivered in-person
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Assessment only (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The investigators adapted two previously validated CBT manuals for use in both Telephone and In-Person groups (the "Personal Health Improvement Program" and Dr. Charles Engel's group treatment for GWI). Treatment included the following standard components of CBT: Didactic or educational material about the causes of GWI and an explanation of how thinking can cause stress ("ABC" model); Assessment of psychological distress and behavioral problems that may be targets of therapeutic intervention (e.g. symptom-related anxiety); Assessment of "thinking errors" that lead to psychological distress and trigger behavioral problems (e.g. catastrophizing); Cognitive restructuring to teach disputing skills or how to correct thinking errors; Cognitive and behavioral homework assignments (e.g. written self-disclosure); Didactic homework assignments (e.g. listen to previous treatment session).
  Arms: In-Person treatment; Telemedicine treatment
Behavioral: Cognitive Behavioral Therapy — This description is the same as the experimental treatment only disseminated in person rather than over the telephone.
  Arms: In-Person treatment; Telemedicine treatment

SUMMARY:
Effective treatments have been developed to ameliorate symptom-related distress and reduce unnecessary healthcare utilization using cognitive-behavioral techniques (CBT) . However there is a major limitation of this treatment is that patients must attend sessions in person. The specific aims of the study are to: (1) Determine the clinical efficacy of Telephone CBT for veterans with GWI who are frequent consumers of ambulatory medical care; (2) Determine whether CBT for veterans with GWI leads to a reduction in the cost of VA health care; and (3) Develop a statistical model of treatment seeking in veterans with GWI who are frequent consumers of ambulatory medical care.

DETAILED DESCRIPTION:
At least as far back as the American Civil War, soldiers have reported nonspecific ailments that could not be attributed to an underlying medical cause. The most frequent symptoms include persistent fatigue, palpitations, headache, muscle or joint pain, disturbed sleep, and cognitive difficulties. Recent epidemiologic studies suggest that war-related syndromes are exceptionally common in deployed personnel and may affect 45% to 60% of returning soldiers. These post-deployment symptoms have substantial consequences that include increased medical visitation, increased physical disability, and increased psychological distress. The number of veterans at risk is likely to increase rather than decrease in the years ahead. In order to address this anticipated increase, new and more efficient treatments for symptom-based illness are urgently needed to augment or replace standard VA care. An effective treatment using cognitive-behavioral techniques (CBT) has been developed to ameliorate symptom-related distress and reduce unnecessary healthcare utilization. Despite convincing evidence of therapeutic efficacy, a major limitation of this treatment is that patients must attend sessions in person. This requirement may undermine the effectiveness of CBT since fewer than half of those who need treatment will attend. A recent trial of CBT for veterans with Gulf War Illness found that only 38% were treatment adherent. Any sudden increase in the number of veterans seeking care could overwhelm the limited resources of a local VA healthcare center. The proposed study will address this important public health problem by testing a cost-effective and innovative strategy for delivering CBT over the phone.

The specific aims of the study are to: (1) Determine the clinical efficacy of Telephone CBT for veterans with GWI who are frequent consumers of ambulatory medical care; (2) Determine whether CBT for veterans with GWI leads to a reduction in the cost of VA health care; and (3) Develop a statistical model of treatment seeking in veterans with GWI who are frequent consumers of ambulatory medical care.

Participation is limited to veterans who satisfy a validated case definition of GWI and whose utilization is at (or above) the 80th percentile. A long-term goal of the proposed research is to make specialized Telephone CBT services widely available to veterans regardless of their geographic location. A previously validated CBT program for GWI has been adapted in consultation with Dr. Charles Engel. The proposed study represents the first randomized (multicenter) trial of Telephone CBT designed to ameliorate GWI and reduce unnecessary reliance on VA health care services. A total of 150 eligible veterans will be assigned to one of three groups: (I) Telephone CBT + Customary Medical Care; (II) In-Person CBT + Customary Medical Care; or (III) Customary Medical Care only.

Revised study procedures were developed and approved by our local IRB. CBT manual was refined and adapted for telephone use. Two postdoctoral fellows were recruited, trained in CBT, and study assessment techniques. A large pool of high utilizing veterans was identified. Of the first 1000 veteran names, 523 were not viable after chart review (outside catchment area; medical rule out; moved; deceased; etc); of 477 remaining 147 were not reachable; 102 declined; 46 were deemed ineligible after initial screening; 49 were eligible and scheduled for psychiatric interview. As of December 2006 a total of 116 veterans have been enrolled in the study and randomized to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Top 20% of medical care utilizers;
* Satisfies criteria for multisymptom illness;
* Enrolled in the New Jersey VA Healthcare System for at least one year

Exclusion Criteria:

* Psychotic disorders;
* Dementia or other cognitive disorders;
* Brain damage;
* Anorexia/other eating disorders;
* Pregnancy;
* Heart failure;
* Cancer;
* Chronic renal insufficiency;
* Severe hepatic disease;
* Active Substance Abuse/Dependence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2008-02-22 (Actual); Study Completion 2008-03-01 (Actual)

PRIMARY OUTCOMES:
Frequency of medical visitation | 12 months

SECONDARY OUTCOMES:
quality of life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mia M Downing, PhD, Principal Investigator — East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ
Locations (1):
- East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey, United States